CLINICAL TRIAL: NCT04136795
Title: Evaluation of the Respiratory Impact of Post-operative Chest Wall Anomalies After Conventional or Minimally Invasive Esophageal Atresia Surgery
Brief Title: Evaluation of the Respiratory Impact After Conventional or Minimally Invasive Esophageal Atresia Surgery
Acronym: RestriMIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut de Recherche en Santé, Environnement et le Travail, France (Other); Filière des Maladies Rares Abdomino-THOraciques : FIMATHO (Unknown)
Responsible Party: Principal Investigator, DENISE JOLIVOT, Dr Françoise Schmitt, University Hospital, Angers
Other Study IDs: 49RC19_0185
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Atresia; Oesophageal Atresia; Restrictive Lung Disease; Chest Wall Anomaly
Keywords: esophageal atresia; thoracoscopy; rib fusion; scoliosis; Respiratory function
MeSH Terms: conditions — Esophageal Atresia; Scoliosis; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional surgery: Patients having had esophageal atresia (type III, long gap excluded) repair by conventional surgery (right thoracotomy) or patients having had minimally invasive surgery converted to thoracotomy between the 1st of january 2008 and the 31st of December 2013 and registered on the national esophageal atresia registry (CRACMO, Lille university hospital)
- Minimally invasive surgery: Patients having had esophageal atresia (type III, long gap excluded) repair through minimally invasive surgery between the 1st of january 2008 and the 31st of December 2013 and registered on the national esophageal atresia registry (CRACMO, Lille university hospital)

SUMMARY:
Right thoracotomy, conventional approach to esophageal atresia repair, leads to up to 60% radiological chest wall sequelae anomalies. The impact of these anomalies on the patient's respiratory function remains unknown. Minimally invasive thoracic surgery considerably reduces this rate.

The primary objective of this study is to assess the occurrence of restrictive lung disease in patients with type III esophageal atresia depending on the type of surgical approach (Conventional or minimally invasive).

The primary endpoint will be he occurrence of restrictive lung disease , objectified by pulmonary function tests (PFTs), carried out according to the current national guidelines (PNDS = protocole national de diagnostic et de soins).

DETAILED DESCRIPTION:
Right thoracotomy, conventional approach to esophageal atresia repair, leads to up to 60% radiological chest wall sequelae anomalies. The impact of these anomalies on the patient's respiratory function remains unknown. Minimally invasive thoracic surgery considerably reduces this rate.

The primary objective of this study is to assess the occurrence of restrictive lung disease in patients with type III esophageal atresia depending on the type of surgical approach (Conventional or minimally invasive).

The primary endpoint will be the occurrence of restrictive lung disease, as assessed by pulmonary function tests (PFTs), carried out according to the current national guidelines (PNDS = protocole national de diagnostic et de soins).

The secondary endpoints will be to measure the severity of the restrictive disease, to look for other respiratory alterations, to correlate radiological chest wall sequelae anomalies with the impact on respiratory function and to look for a causal relationship between the surgical technique used and the respiratory impact.

The methodology used will be a retrospective non interventional study on the cohort of patients included in the national esophageal atresia registry (CRACMO, Lille University Hospital) between the 1st of january 2008 and the 31st of December 2013.

All the patients included in the national esophageal atresia registry (CRACMO) having had an operation for type III esophageal atresia (long gap esophageal atresia excluded), as defined by the Ladd Classification, will be included in this study.

The exclusion criterion will be patients lost to follow up or deceased, patients having had no pulmonary function tests (PFTs) or no thoracic X-Ray during the first 6 to 9 years of follow up and patients having had thoracic surgery before the esophageal atresia repair.

The number of patients expected in the national esophageal atresia registry over the 6 years excedes 500. The number of thoracoscopy repairs should be about 50.

This study should allow us to determine if minimally invasive surgery is beneficial on mid-term respiratory function in children, related to possible post-operative chest wall sequelae.

The results obtained from this study should lead to recommendations concerning the surgical approach to esophageal atresia repair to improve the prognosis of chest wall anomalies and respiratory function in these patients. It should also help to identify patient subgroups which would benefit from a reinforced respiratory follow up. This could then lead to a hospital clinical research program (PHRC)

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the national esophageal atresia registry (CRACMO)
* Operation for type III esophageal atresia (Ladd classification)
* Between 01/01/2008 and 31/12/2013.

Exclusion Criteria:

* Long gap esophageal atresia
* Patients lost to follow up
* Deceased
* No PFTs or X-rays between 6 and 9 years of follow up
* Patients having had thoracic surgery before the esophageal atresia repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients included in the national esophageal atresia registry (CRACMO) having had an operation for type III esophageal atresia, as defined by the Ladd classification between 01/01/2008 and 31/12/2013 and being followed up with thoracic X-rays and PFTs.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To assess the occurrence of restrictive lung disease in patients with type III esophageal atresia depending on the type of surgical approach (Conventional or minimally invasive). | 6 to 9 years of age.
  Objectified by pulmonary function tests (PFTs), carried out according to the current national guidelines. Restrictive lung disease defined by: FEV1/FVC ratio > -1.64 Z-score and CVF < -1.64 Z-score according to ATS/ERS-GLI (American Thoracic Society & European Respiratory Society - Global Lungs Initiative) recommendations.

SECONDARY OUTCOMES:
Severity of restrictive lung disease | 6 to 9 years of age
  Depending on Z-score value
Assesse the occurrence of obstructive or mixed lung disease | 6 to 9 years
  Objectified by pulmonary function tests (PFTs), carried out according to the current national guidelines. Mixed lung disease defined by: FEV1/FVC ratio < -1.64 Z-score and CVF < -1.64 Z-score and obstructive lung disease
Mortality rate | Time of surgery to 6 to 9 years consultation
  Percentage of mortality in each group, cause of death linked directly to surgery or not
Percentage of post-operative complications depending on the type of surgery | Time of surgery to 6 to 9 years consultation
  Bleeding, infection, anastomotic stenosis, anastomotic leak
Chest wall anomalies detected on thoracic X-rays | 6 to 9 years of age
  Hemivertebra, rib fusion, intercostal abnormalities, scoliosis
Correlation between post-operative chest wall anomalies and restrictive lung disease | 6 to 9 years of age
  In each group, comparison of the percentage of chest wall anomalies detected on the X-rays and the percentage of restrictive lung disease cases

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Schmitt, MD, PhD, Principal Investigator — University Hospital of Angers
Locations (1):
- CRACMO - centre de référence des atrésies de l'oesophage, Lille, France

REFERENCES:
- [Result] Bastard F, Bonnard A, Rousseau V, Gelas T, Michaud L, Irtan S, Piolat C, Ranke-Chretien A, Becmeur F, Dariel A, Lamireau T, Petit T, Fouquet V, Le Mandat A, Lefebvre F, Allal H, Borgnon J, Boubnova J, Habonimana E, Panait N, Buisson P, Margaryan M, Michel JL, Gaudin J, Lardy H, Auber F, Borderon C, De Vries P, Jaby O, Fourcade L, Lecompte JF, Tolg C, Delorme B, Schmitt F, Podevin G. Thoracic skeletal anomalies following surgical treatment of esophageal atresia. Lessons from a national cohort. J Pediatr Surg. 2018 Apr;53(4):605-609. doi: 10.1016/j.jpedsurg.2017.07.013. Epub 2017 Jul 21. PMID 28778692
- [Derived] Chansou MA, Sfeir R, Bonnard A, Rousseau V, Gelas T, Guinot A, Habonimana E, Micheau P, Ranke A, Talon I, Irtan S, Lamireau T, Rabattu PY, Elbaz F, Kalfa N, Panait N, Fouquet V, Lardy H, Scalabre A, Buisson P, Margaryan M, Auber F, Grosos C, Borderon C, Tolg C, Goulin J, Podevin G, Gottrand F, Schmitt F. Retrospective case-control study of nutritional and respiratory status in children with type III esophageal atresia. J Pediatr Gastroenterol Nutr. 2026 Jan;82(1):184-193. doi: 10.1002/jpn3.70238. Epub 2025 Oct 17. PMID 41104659